CLINICAL TRIAL: NCT03662945
Title: Mobile Geriatric Teams: A Cost-effective Way of Improving Patient Safety and Reducing Traditional Healthcare Utilization Among the Frail Elderly?
Brief Title: Mobile Geriatric Teams: Patient Safety and Healthcare Utilization
Acronym: MGT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jonkoping University (Other)
Collaborators: Region Jönköping County (Other Government)
Responsible Party: Principal Investigator, Sofi Fristedt, Ph D, Senior lecturer, Jonkoping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MGT FUTURUM-521121
Record Dates: First submitted 2018-08-10; First posted 2018-09-10 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Frail Elderly Syndrome

STUDY DESIGN:
Intervention Model Description: 1 intervention group and 1 control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Mobile Geriatric Team intervention including physicians and nurses with the aim of developing person-centered, safe, sustainable and coordinated care plans. These care plans are developed in collaboration with the patient, his/her relatives and staff from the municipality. Among the main ambitions of this concept are improved communication flows between patients, their relatives and healthcare providers in combination with the delivery of medical as well as care measures. Other ambitions are to avoid unnecessary traditional healthcare utilization in the form of inpatient care and EMR visits, for example.
  Interventions: Other: Mobile Geriatric Team intervention
- Control group (No Intervention): Standard care including primary care units, home care and home help.

INTERVENTIONS:
Other: Mobile Geriatric Team intervention — Person-centred intervention based on Comprehensive Geriatric Assessment
  Arms: Intervention group

SUMMARY:
Objective To perform a prospective, controlled and randomized evaluation of the effectiveness of Mobile Geriatric Teams (MGT).

Method Community-dwelling, frail elderly people were randomized to intervention group (n=31, mean age 84) and control group (n=31, mean age 86). Two-year retrospective data and prospective one-year follow up, were analyzed using non-parametric and difference-in-difference (DiD) analyses. Qualitative interviews, were analyzed using content analysis.

DETAILED DESCRIPTION:
Method The current study was conducted through a randomized control trial (RCT), upon approval from the Regional Ethical Committee in Linköping, Dnr 2014/371-31. The study context was an MGT, initiated in 2013 and originated from a hospital serving approximately 149,000 inhabitants in Southern Sweden.

Participants The inclusion criteria for this trial were the "frail elderly" defined as: community-dwelling persons aged > 75 years, having more than three chronic diagnoses and prescribed six or more pharmaceutical drugs for continuous use and with at least three hospital stays (> 24 hours in hospital) during the last six months. Since these criteria were broad in order to capture relevant individuals, but also likely to generate persons of no relevance to the MGT intervention, identification of the study sample was conducted in three steps, in turn, repeated in three waves.

In the first step, a nurse with special training in identifying populations by filtered searches in digital patient records identified 449 individuals in an initial search (March 2015). Another 75 individuals were identified in a second search wave (May 2015) and another 157 individuals in a third search wave (September 2015).

In the second step, a nurse with geriatric competence checked the patient records of all individuals. Deceased persons or persons who had moved to a nursing home since the initial search were excluded. Patients with repeated hospital admissions due to surgery (without multi-morbidity) or patients admitted for palliative care were also excluded from the sample. Thirdly and finally for all waves, a nurse with clinical experience of MGT re-evaluated each of the previous searches in order to exclude individuals that the MGT would not consider for inclusion, since they were likely to not benefit from the MGT measures.

The final recruitment of participants from the above-described filtering resulted in 66 potential participants from the first search, 34 from the second search and 41 from the third search. These were randomized, as shown in Figure 2, to an intervention group and a control group, comprising 31 participants each and an administrative control group, not contacted or followed in the present trial. The initial intention was only to observe the administrative control group data from health and social care registers, but for (the purpose of) the present study this was never done.

The potential participants in control group were contacted via telephone and the aim of the study was communicated both orally and in writing before the study commenced. Persons sampled to the intervention group, were first informed on the intervention and made their decision on whether to take part in that or not, before being informed (orally and in writing) about the study. All persons who agreed to the MGT-intervention also gave their consent to be part of the study (intervention group). All participants were given the chance to ask questions before their informed consent.

Intervention The intervention started with a home visit. During the first visit, a comprehensive geriatric assessment (CGA) (Ellis et al., 2011) was conducted, together with a pharmaceutical review. Based on this, a person-centered and coordinated as well as (hopefully) sustainable care plan was developed by the MGT, in collaboration with the patient, his/her relatives and the homecare staff. Overall medical responsibility for the patient was temporarily transferred to the MGT physician from primary care during the intervention period. The initial intention was for this to last for 15 weeks but based on early experience the time limit was removed, since it was considered inadequate to break the continuity, and since the primary care units would have problems keeping the same level of continuity of service. Thus, the MGT "retained" the patient as long as was considered necessary. The result of this change was that the enrollment from the MGT was not withdrawn unless the participant moved to a nursing home, re-gained stable health, or died, and, in individual cases, at the patient's request. If patients required palliative care, the MGT remained responsible but consulted an already-existing external palliative team when necessary. After the initial visit, patients were free to contact the MGT during office hours (08.00-17.00) and were referred to home care or hospital outside these hours. Additional visits from nurses, physicians or the whole team were often scheduled on regular basis, but were also possible to arrange at short notice, i.e. on the same day.

Fully operative and in full-time equivalents, the MGT team comprised 1.95 physicians and 3.2 nurses during 2016. They cared for a stock of around 95-100 patients, matching their capacity. Based on presumed discharges, they had the capacity to register an estimated 200 patients annually. The team had access to external equipment, for example, cars and mobile electronic patient records with updated lists of medication and all other information about the patient in the in-hospital patient records. The dictation of measures was performed via laptops. The main costs of the MGT initiative comprise personnel and, in total, this amounts to around Swedish Krona (SEK) 3.7 million annually (around 430,000 United States Dollars based on an exchange rate of 8.56 SEK, provided by the Swedish Central Bank for 2016), including salaries, payroll taxes and social charges. Hence, the average annual personnel cost per patient year is around SEK 37,000 SEK (or SEK 18,500 per estimated new annual registration in fully functional mode). To put this in perspective, the cost of traditional care has been calculated by the county council at, for example, SEK 6,500 for inpatient geriatric care days and SEK 1,600 SEK Emergency Room (EMR) visits. Hence, the MGT initiative must have apparent effects on traditional health care utilization in order to reach economic break-even and be self-financed.

Taking the estimated capacity of taking care of up to 200 patients annually literally implies that the traditional care consumption of the average MGT patient has to be reduced annually by about 2.85 care days or 11.6 EMR visits (or a combination of both) in order to reach break-even and be self-financed.

Instruments and variables Data collection was conducted retrospectively via comprehensive county council and municipal administrative registers covering all inhabitants regarding healthcare consumption, home care and home help given to participants as shown in Table 1.

Healthcare consumption was measured via the number of EMR visits, number of hospital admissions, number of days admitted to hospital, outpatient visits to hospital. Primary care consumption was measured via number of visits to a) physicians and b) nurses. Note that care given by, and contact with, the MGT team were not included in any of these measurements. Moreover, participants were contacted and, during a home visit, data on performance in Activities in Daily Living (ADL) (bathing, dressing/undressing, toileting, transfers, continence, eating) were collected through the Katz ADL index (Brorsson & Hulter Åsberg, 1984). In this index, ADL is measured along a seven-point scale (i.e. 1=independent in all activities, 2=dependent in one activity, 3=dependent in bathing and one additional activity, 4=dependent in bathing, dressing/undressing and one additional activity, 5=dependent in bathing, dressing/undressing, toileting and one additional activity, 6=dependent in bathing, dressing/undressing, toileting, transfers and one toileting activity, 7=dependent in all six activities. Moreover, cognitive function was screened using Mini-Mental State Examination (MMSE), ranging from 0-30 points (Folstein, Robins, & Helzer, 1983).

Both groups were interviewed following a structured guide that covered subjective health, subjective safety and security, and their experiences of care given by hospital units or primary units, as well as home help and home care. At inclusion, participants and relatives in the intervention group were asked for their expectations of the coming measures from MGT. Questions regarding experiences of the performed measures were asked and documented 15 weeks later. All face-to-face data collections were done by the project manager (first author) or an (the same) research assistant (RN).

Analysis Variation in healthcare utilization pre- and post the MGT intervention was compared for the control and intervention group, respectively, as well as between groups pre- and post-intervention via two-sample Wilcoxon rank-sum (Mann-Whitney) tests. In order to discern whether the MGT treatment had any causal effects on healthcare utilization, the data were assessed via a difference-in-difference (DiD) analysis, in which the change in utilization following the introduction of MGT in the treatment group was compared to the corresponding development of the unaffected control group during the same time frame. The DiD analysis is estimated via linear regression and the reported significance values obtained using robust standard errors.

The qualitative interviews were transcribed verbatim. Meaning units were identified, condensed and coded. Codes were abstracted into two categories based on similarities and given content-describing names.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria for this trial were the "frail elderly" defined as:

* community-dwelling persons aged > 75 years,
* having more than three chronic diagnoses,
* prescribed six or more pharmaceutical drugs for continuous use and
* with at least three hospital stays (> 24 hours in hospital) during the last six months.

Since these criteria were broad in order to capture relevant individuals, but also likely to generate persons of no relevance to the MGT intervention, identification of the study sample was conducted in three steps, in turn, repeated in three waves.

Exclusion Criteria:

* Persons not able to take part in qualitative interviews

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2015-12-20 (Actual); Study Completion 2015-12-20 (Actual)

PRIMARY OUTCOMES:
Health care utilization including EMR, hospital admissions, care days, out patient hospital or primary care | Change from 1 year before inclusion to 1 year follow up
  No. of EMR visits, Out patient visits to hospital, Hospital admissions, Care days, Primary care visits

SECONDARY OUTCOMES:
Health care utilization including EMR, hospital admissions, care days, out patient hospital or primary care | Change from 2 year before inclusion to 1 year follow up
  No. of EMR visits, Out patient visits to hospital, Hospital admissions, Care days, Primary care visits
Health care utilization including EMR, hospital admissions, care days, out patient hospital or primary care | Change from inclusion to 3 year follow up
  No. of EMR visits, Out patient visits to hospital, Hospital admissions, Care days, Primary care visits

OTHER OUTCOMES:
Patient and next-of-kin satisfaction assessed by Qualitative interviews | Changes from inclusion to 15 week follow-up
  Qualitative interviews on patient safety and patient /next-of-kin satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Sofi Fristedt, Ph D, Principal Investigator — Jonkoping University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fristedt S, Nystedt P, Skogar O. Mobile Geriatric Teams - A Cost-Effective Way Of Improving Patient Safety And Reducing Traditional Healthcare Utilization Among The Frail Elderly? A Randomized Controlled Trial. Clin Interv Aging. 2019 Nov 5;14:1911-1924. doi: 10.2147/CIA.S208388. eCollection 2019. PMID 31806947